CLINICAL TRIAL: NCT03442790
Title: Agitated Saline Versus Chest X-ray for Determination of Correct Position of Central Venous Catheter: a Non-inferiority Study
Brief Title: Agitated Saline Versus CXR Confirmation of Central Venous Lines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Dr. Achyut Sharma, MD Anesthesia and Intensive Care, Nepal Mediciti Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NepalMediciti
Record Dates: First submitted 2018-02-10; First posted 2018-02-22 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Central Venous Catheterization; Exposure to X-Rays
Keywords: CVC confirmation; Agitated Saline; CXR
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants will not have any knowledge of the intervention and the investigator who is doing the ultrasound confirmation will not have access to the results of the chest x-ray confirmation until the end of the study period when all the data is analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agitated Saline Method (Experimental): The proper placement of the central venous line will be confirmed using agitated saline under ultrasound vision
  Interventions: Procedure: Agitated Saline Method; Procedure: chest x-ray
- Chest X-Ray Confirmation (Active Comparator): The proper placement of the central venous line will be compared with chest x-ray obtained in supine position after central line placement
  Interventions: Procedure: Agitated Saline Method; Procedure: chest x-ray

INTERVENTIONS:
Procedure: Agitated Saline Method — All patients in the study who have undergone a central venous line placement will undergo a confirmation of the accurate or inaccurate placement of central venous lines using agitated saline under ultrasound vision.
  Other Names: bubble confirmation; contrast enhanced confirmation
Procedure: chest x-ray — All patients in the study who have undergone a central venous line placement will undergo a confirmation of the accurate or inaccurate placement of central venous lines using chest x-ray obtained in supine position as an active comparator
  Other Names: CXR; supine x-ray

SUMMARY:
Central venous lines insertion are common procedures these days. CVL placed under USG guidance have high success rates and low complications even in developing country settings. However, the investigators still have to rely on chest x-ray (CXR) to confirm the correct placement of central venous lines as a gold standard method. This might be time consuming and may cause delay in initiation of treatment. In some cases, as in operating room, the treatment is started even before confirmation by CXR. Ultrasound has ability to localize the tip of the catheter at the superior venacava- right atrium junction using agitated saline and the appearance of contrast within 2 seconds in right atrium. However, this technique is rarely used. The investigators, therefore, designed the trial to study whether confirmation of tip of CVL by ultrasound is non-inferior to the CXR confirmation.

DETAILED DESCRIPTION:
Central venous lines (CVL) are placed in various in-hospital settings like operation theaters, emergency departments, oncology departments, and intensive care units for various purposes. Like any invasive procedures, placement of central lines is invariably associated with certain risks of inadvertent complications which are often life-threatening which occur because of the intricacy of the structures around the vascular access site like pleura, arteries, nerves, heart, etc. Measures such as landmark guidance, electrocardiographic guidance, fluoroscopy/C-arm-guided, and recently ultrasound image guidance have been in place to prevent and/or minimize the occurrence of such complications. Although the incidence of such complications have decreased considerably4, the rates have not reached the nadir.

Failure of confirmation of the correct placement of a CVL can have serious consequences. The consequences of an inadvertently misplaced catheter are grave for the patient be it the failure to elicit the vasopressor effect, unnecessary delay in starting of caustic substances like hypertonic fluids, parenteral nutrition, concentrated agents, etc., these will ultimately increase the morbidity and mortality. Thus, it becomes imperative that we confirm the accurate placement of CVL before infusing anything through these lines.

The confirmation of accurate placement of CVL is usually done by performing a post-procedure chest x-ray (CXR) which is done at the point of care if possible like in ICU or after shifting of patient to a post-operative ward in an operation theater setup. The most important constraint in obtaining CXR after CVL placement is the considerable amount of time it takes before a film is obtained even in center where there is a dedicated portable CXR for that purpose. For CVL placed in the operating theater, it is not always possible to do a portable CXR immediately after the procedure and at many times we have to immediately start infusion/medications through it even before confirmation of their proper placement. Secondly the very well-known problem of radiation hazard is a potential deterrent to the use of CXR each time a CVL is placed. When a large volume ICU is compared, the risk of radiation is inadvertently extended to all of the patients even though lines are placed in some. The hazard of the radiation to the ICU and ED staffs is always a concern considering the difficulty they face in escaping the hazard when they are taking care of sick patients. Thirdly, it is difficult to obtain an accurate CXR film in critical care unit setups where the patient are sometimes unable to hold breaths at inspiration (for the proper x-ray film) and the film so obtained may not be reliable enough to read. Fourthly, the overall costs in obtaining CXR for each and every single central lines placed will add to the overall healthcare costs at a time when the investigators are looking for reasons to cut down on health expenses.

Considering the fact that these lines are placed under ultrasound guidance, the rate of inadvertent complications are very few. But subjecting every single individual to an x-ray cannot always be justified. Nevertheless, this is not to say that central lines should not be confirmed for their proper placement, but certainly there is an imminent need of a simple, reliable, and more cost effective alternative to CXR. The very same ultrasound machine at point of care can be utilized for this purpose addressing most of the limitations of the CXR.

With simple, directed teaching it is possible for anyone with basic knowledge in ultrasound to do a focused point of care ultrasound to evaluate the accurate placement of CVL. This simple approach has several potential benefits. The first one being the saving of precious post-procedure time that is lost in obtaining a chest x-ray. The potential radiation hazard due to CXR is virtually eliminated. The same ultrasound can also be utilized for scanning the thorax to exclude pneumothorax and hemothorax and avoid potential delay in their management. If the sensitivity and specificity of ultrasound in accurately delineating the position of CVL is comparable to the chest x-ray, then obtaining of chest x-ray for confirmation can virtually be eliminated.

Although, it is possible to see the intravascularly placed CVL by scanning the respective vessel and visualizing the acoustic shadow in transverse axis and following the same in longitudinal axis, there is a limitation to the extent these lines can be followed to. The user who is usually positioned just above the head has access to scan the neck veins and follow the vessels until the bony structures like clavicle and ribs limit further interpretation unless we are using a transesophageal echocardiography. Thus, experts have devised a noble technique of using agitated saline as contrast agent to check the accurate location of central line. When performed properly, the contrast agent which is injected through the distal most port of central line will create a wave of microbubbles appearing to enter the right atrium from superior venacava and the relative time it takes for these bubbles to appear help interpret the position of CVL with a relatively high degree of sensitivity and specificity. This simple yet effective method is not expected to take a long time to perform. However, not all the studies thus performed so far have been consistent in obtaining a conclusive evidence of its effectivity and sensitivity. Most of the studies done till date have been relatively underpowered by a small sample size to draw a major conclusion as to justify the use of ultrasound in detection of CVL placement. This very finding dictates the necessity of conducting even more studies in diverse groups of population before a concrete conclusion is drawn. Unlike previous studies where the ultrasound was compared as an absolute method to completely replace the CXR in confirmation of CVL which still seems to be far-fetched idea, the investigators seek to see that ultrasound guided agitated saline method of confirmation is not inferior to chest x-ray in confirming or refuting the accurate placement of CVL. By this study, the investigators do not at all seek to completely eliminate chest x-ray in confirmation of CVL but at least make an interpretation by using appropriate tests that ultrasound has the potential to be effective in decreasing the necessity of CXR in post-CVL insertion confirmation. The investigators believe that rather than subjecting every single person to radiation hazard after CVL, it is justifiable to obtain CXR only in those cases where there is confirmatory dilemma with agitated saline. Till date, there are also no specific guides to accurately predict the length at which the CVL should be fixed at skin before any form of confirmation can be done. The investigators assume that with this study, they will be able to better able to tell what is the most appropriate length of CVL fixing which can be extended to other patients of similar population group. Also, the investigators presume that it is possible to virtually eliminate a large numbers of unnecessary x-rays including all of their hazards and also cut down the healthcare costs. The investigators also believe that in the due course of time, with this and other similar and sufficiently powered studies, it will be possible to draw a firm conclusion and use ultrasound as an effective tool for its varied purposes in intensive care and emergency settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years admitted to ICU or presenting to operation theater for surgical procedures
2. Patients with indications for above the diaphragm CVL placement
3. All above the diaphragm central venous lines placed under ultrasound guidance.

Exclusion Criteria:

1. Age <18 years
2. Pregnant patients
3. Patients with moderate and severe RV dysfunction
4. Patient with moderate and severe tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of central line placement | 7 months
  1. To compare the accuracy of ultrasound guided agitated saline confirmation and chest x-ray confirmation of central venous line position

SECONDARY OUTCOMES:
Compare the time required for confirmation | 7 months
  To compare the time required for ultrasound guided agitated saline confirmation and chest x-ray confirmation of central venous line position
Accuracy of malposition detection | 7 months
  To compare the accuracy of detection of central venous line malposition

CONTACTS AND LOCATIONS:
Overall Officials: Achyut Sharma, MD, Principal Investigator — Nepal Mediciti Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mulvany SA, Mcconkey C, Allen S. An Audit of Central Venous Line Insertion, the use of Ultrasound Guidance and the Incidence of Carotid Artery Puncture. Int J Perioper Ultrasound Appl Technol Int J Periop Ultrasound Appl Technol. 2012;1(33):99-101.
- [Background] Joshi AM, Bhosale GP, Parikh GP, Shah VR. Optimal positioning of right-sided internal jugular venous catheters: comparison of intra-atrial electrocardiography versus Peres' formula. Indian J Crit Care Med. 2008 Jan;12(1):10-4. doi: 10.4103/0972-5229.40943. PMID 19826584
- [Background] Gebauer B, Teichgraber UM, Werk M, Beck A, Wagner HJ. Sonographically guided venous puncture and fluoroscopically guided placement of tunneled, large-bore central venous catheters for bone marrow transplantation-high success rates and low complication rates. Support Care Cancer. 2008 Aug;16(8):897-904. doi: 10.1007/s00520-007-0378-9. Epub 2008 Jan 16. PMID 18197436
- [Background] Palepu GB, Deven J, Subrahmanyam M, Mohan S. Impact of ultrasonography on central venous catheter insertion in intensive care. Indian J Radiol Imaging. 2009 Jul-Sep;19(3):191-8. doi: 10.4103/0971-3026.54877. PMID 19881083
- [Background] Pikwer A, Baath L, Davidson B, Perstoft I, Akeson J. The incidence and risk of central venous catheter malpositioning: a prospective cohort study in 1619 patients. Anaesth Intensive Care. 2008 Jan;36(1):30-7. doi: 10.1177/0310057X0803600106. PMID 18326129
- [Background] Matsushima K, Frankel HL. Bedside ultrasound can safely eliminate the need for chest radiographs after central venous catheter placement: CVC sono in the surgical ICU (SICU). J Surg Res. 2010 Sep;163(1):155-61. doi: 10.1016/j.jss.2010.04.020. Epub 2010 May 11. PMID 20599208
- [Background] Xie Z, Liao X, Kang Y, Zhang J, Jia L. Radiation Exposure to Staff in Intensive Care Unit with Portable CT Scanner. Biomed Res Int. 2016;2016:5656480. doi: 10.1155/2016/5656480. Epub 2016 Jul 31. PMID 27556036
- [Background] Andropoulos DB, Stayer SA, Bent ST, Campos CJ, Bezold LI, Alvarez M, Fraser CD. A controlled study of transesophageal echocardiography to guide central venous catheter placement in congenital heart surgery patients. Anesth Analg. 1999 Jul;89(1):65-70. doi: 10.1097/00000539-199907000-00012. PMID 10389780
- [Background] Cortellaro F, Mellace L, Paglia S, Costantino G, Sher S, Coen D. Contrast enhanced ultrasound vs chest x-ray to determine correct central venous catheter position. Am J Emerg Med. 2014 Jan;32(1):78-81. doi: 10.1016/j.ajem.2013.10.001. Epub 2013 Oct 9. PMID 24184012
- [Background] Rezayat T, Stowell JR, Kendall JL, Turner E, Fox JC, Barjaktarevic I. Ultrasound-Guided Cannulation: Time to Bring Subclavian Central Lines Back. West J Emerg Med. 2016 Mar;17(2):216-21. doi: 10.5811/westjem.2016.1.29462. Epub 2016 Mar 2. PMID 26973755